CLINICAL TRIAL: NCT00335569
Title: A Prospective, Randomized, Controlled Clinical Study on the Assessment of Tolerance and Clinical Equivalence of hCG- IBSA (IBSA) Versus Ovitrelle (Serono), Both Administered Sub-cutaneously in Women Undergoing in Vitro Fertilization (IVF).
Brief Title: Clinical Tolerance and Equivalence of hCG-IBSA vs Recombinant Human Chorionic Gonadotrophin in Women Undergoing In Vitro Fertilisation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04CH/HCG02
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Infertility
Keywords: Infertility, sterility, hCG, IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hCG-IBSA

SUMMARY:
The purpose of the study is to evaluate the clinical equivalence and the general tolerability of two different subcutaneous hCG preparations (hCG-IBSA, IBSA vs Ovitrelle, Serono) when administered to patients undergoing IVF.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, investigator blind, parallel group, active control, phase III clinical trial. Patients meeting the eligibility requirements of the study will be randomly assigned to receive either the test drug (hCG-IBSA, IBSA) or the reference drug (Ovitrelle, Serono). Investigators will be blinded by not allowing them to have any contact with the study medications (supplied in boxes labeled in a manner that does not reveal the content of the boxes), and requesting that patients do not make any statements to the investigator that might indicate the treatment to which they were assigned. Equivalence testing with regard to the primary outcome variable will establish whether the two treatments are indeed similarly effective.

ELIGIBILITY:
Inclusion Criteria:

* >/=18 and < 40 years old;
* BMI between 18 and 30 kg/m2;
* less than 3 previous completed cycles;
* both ovaries present;
* regular menstrual cycle of 25-35 days;
* infertility attributable to a tubal factor, American Fertility Society grade I or II endometriosis, male factor or unexplained factor.
* within 12 months of the beginning of the study, uterine cavity consistent with expected normal function as assessed through hysterosalpingogram, sonohystrogram or hysteroscopic examination;
* basal FSH level less than 10 IU/L;
* criteria for hCG administration fulfilled (at least 2 follicles with a diameter of 16 mm or more, with acceptable serum E2 concentration).
* a male partner with semen analysis within the past 6 months showing acceptable values of seminal parameters, defined as > 3x10 exp 6 spermatozoa/ml;
* qualified to receive 150 - 300 IU FSH as starting dose.

Exclusion Criteria:

* age < 18 and > o = 40 years;
* primary ovarian failure or women known as poor responders (i.e. requiring more than 300 IU of FSH as a starting dose in previous treatment cycles or having less than 3 oocytes retrieved, or with an E2 serum concentration < 3'000 pmol/L);
* ovarian cysts > 20 mm, or enlargement not due to polycystic ovarian syndrome;
* patients affected by pathologies associated with any contraindication of being pregnant;
* hypersensitivity to the study medication;
* any bleeding since stimulation;
* uncontrolled thyroid or adrenal dysfunction;
* neoplasias;
* severe impairment of the renal and/or hepatic functions;
* use of concomitant medication that might interfere with study evaluations (e.g. nonstudy hormonal medications, prostaglandin inhibitors, psychotropic agents);
* more than 18 days of FSH stimulation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2005-08; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Total number of oocytes retrieved per patient who received hCG

SECONDARY OUTCOMES:
Number of patients who received hCG with at least one oocyte retrieved, 2PN fertilized oocytes,
2PN or cleaved embryos, implantation rate per embryo transferred; Serum P and hCG concentration on the days of oocyte retrieval, on day of embryo transfer and on day 5-8 post-hCG;
Implantation rate;Pregnancy rate.
Adverse Events | from day 1 to 35 +/- 7 days after oocytes retrieval
  Adverse events were monitored and collected during all the study period
Incidence of moderate or severe OHSS | From the day of hCG injection until 35 +/- 7 days after oocyte retrieval
  The incidence moderate or severe of OHSS will be assessed in both treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Ziegler, Prof., Principal Investigator — Départements de Gynécologie/Obstétrique et de Pédiatrie
Locations (4):
- Switzerland (4):
  - Department of Gynecology and Obstetrics Universitätfrauenklinik, Basel
  - 4. Department of Gynecology and Obstetrics Frauenklinik, InselspitalEffingerstrasse 102, Bern
  - Department of Gynecology and ObstetricsUniversity Hospital, Geneva
  - 3. Maternity CHUV - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Background] Pierce JG, Parsons TF. Glycoprotein hormones: structure and function. Annu Rev Biochem. 1981;50:465-95. doi: 10.1146/annurev.bi.50.070181.002341. No abstract available. PMID 6267989
- [Background] Johnsen SG. A study of human testicular function by the use of human menopausal gonadotrophin and of human chorionic gonadotrophin in male hypogonadotrophic eunuchoidism and infantilism. Acta Endocrinol (Copenh). 1966 Oct;53(2):315-41. doi: 10.1530/acta.0.0530315. No abstract available. PMID 6012569
- [Background] Forest MG, David M, Lecoq A, Jeune M, Bertrans J. Kinetics of the HCG-induced steroidogenic response of the human testis. III. Studies in children of the plasma levels of testosterone and HCG: rationale for testicular stimulation test. Pediatr Res. 1980 Jun;14(6):819-24. doi: 10.1203/00006450-198006000-00009. PMID 6105640
- [Background] GEMZELL C. INDUCTION OF OVULATION WITH HUMAN GONADOTROPINS. Recent Prog Horm Res. 1965;21:179-204. No abstract available. PMID 14321057
- [Background] Fleischer AC. Transabdominal and transvaginal sonography of ovarian masses. Clin Obstet Gynecol. 1991 Jun;34(2):433-42. doi: 10.1097/00003081-199106000-00027. PMID 1868645
- [Background] Vermesh M, Kletzky OA. Follicle-stimulating hormone is the main determinant of follicular recruitment and development in ovulation induction with human menopausal gonadotropin. Am J Obstet Gynecol. 1987 Dec;157(6):1397-402. doi: 10.1016/s0002-9378(87)80231-4. PMID 3122575
- [Background] Brown JB, Evans JH, Adey FD, Taft HP, Townsend L. Factors involved in the induction of fertile ovulation with human gonadotrophins. J Obstet Gynaecol Br Commonw. 1969 Apr;76(4):289-307. doi: 10.1111/j.1471-0528.1969.tb05837.x. No abstract available. PMID 5778792
- [Background] Venturoli S, Paradisi R, Fabbri R, Magrini O, Porcu E, Flamigni C. Comparison between human urinary follicle-stimulating hormone and human menopausal gonadotropin treatment in polycystic ovary. Obstet Gynecol. 1984 Jan;63(1):6-11. PMID 6419189
- [Background] Abdalla HI, Ah-Moye M, Brinsden P, Howe DL, Okonofua F, Craft I. The effect of the dose of human chorionic gonadotropin and the type of gonadotropin stimulation on oocyte recovery rates in an in vitro fertilization program. Fertil Steril. 1987 Dec;48(6):958-63. doi: 10.1016/s0015-0282(16)59591-0. PMID 3119376
- [Background] Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E. Ovarian hyperstimulation syndrome: an update review. Obstet Gynecol Surv. 1989 Jun;44(6):430-40. doi: 10.1097/00006254-198906000-00004. No abstract available. PMID 2660037
- [Background] Hauschke D, Kieser M, Diletti E, Burke M. Sample size determination for proving equivalence based on the ratio of two means for normally distributed data. Stat Med. 1999 Jan 15;18(1):93-105. doi: 10.1002/(sici)1097-0258(19990115)18:13.0.co;2-8. PMID 9990695
- [Derived] Bellavia M, de Geyter C, Streuli I, Ibecheole V, Birkhauser MH, Cometti BP, de Ziegler D. Randomized controlled trial comparing highly purified (HP-hCG) and recombinant hCG (r-hCG) for triggering ovulation in ART. Gynecol Endocrinol. 2013 Feb;29(2):93-7. doi: 10.3109/09513590.2012.730577. Epub 2012 Nov 2. PMID 23116325